CLINICAL TRIAL: NCT05443386
Title: Emergency Surgery for Colon Diseases in Elderly Patients. Analysis of Complications, and Postoperative Course
Brief Title: Colorectal Emergencies in Elderly Patients.
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Mario Pacilli, Principal Investigator, University of Foggia
Other Study IDs: UFoggia1
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Emergency Colorectal Surgery in Ultra 80 Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colorectal surgery — we have included several types of colorectal surgery procedures, in emergency conditions

SUMMARY:
Colon diseases can turn in a clinical emergency with the onset of some important complications. Some critical conditions are more common in aged patients because they are more frails. The aim of this study is to examine ultra 80 patients, undergoing emergency colorectal surgery, evaluating the aspects associated with post-operative complications and other problems in the short term.

From November 2020 to February 2022 we have included 32 consecutive patients older than 80 undergoing emergency surgery due to colon diseases. We have collected and analysed all demographic, and operative data and then applied CR-POSSUM score and correlated with postoperative hospital stay and the onset of postoperative complications according to Clavien Dindo classification.

Postoperative factors were selectively evaluated based on the clinical scenario and different colic pathologies. There was no statistically significant differences, in terms of postoperative hospital stay, postoperative complications, reoperation rate and 30-day mortality. The number of cases of blood transfusions was significant, more numerous in case of intestinal perforation and bleeding cases. The value of Operative Severity Score in the Bowel Perforations, was significantly higher.

The use of a score to stratify the risk is a useful tool especially in elderly patients to undergo emergency surgery. The CR-POSSUM score was important for predicting morbidity in our study. Emergency manifestations of colon diseases in the elderly show higher morbidity and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* age older than eighty
* emergency conditions

Exclusion Criteria:

* trauma cases

Min Age: 80 Years | Sex: All
Age Groups: Older Adult
Study Population: patients older than 80 undergoing emergency surgery (within 24 hours) due to colon diseases were included in this retrospective study
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
postoperative hospital stay | 30 days

SECONDARY OUTCOMES:
postoperative complications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Di Foggia, Foggia, Italy

DOCUMENTS (1):
  • Study Protocol (2022-06-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT05443386/Prot_000.pdf